CLINICAL TRIAL: NCT04158609
Title: Assessment of the Relationship Between Delivery Route, Umbilical Cord pH and Fetal Complications With Doppler Parameters Measured Prior to Induction of Labor at Term Pregnancies.
Brief Title: Relationship Between Delivery Route and Fetal Complications With Doppler Indices and CPR Parameters
Acronym: Doppler
Status: Completed | Type: Observational
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Özkan Özdamar, M.D., Principal Investigator, Clinical Investigator of OB&GYN, Istanbul Medeniyet University
Other Study IDs: 2018/0473
Record Dates: First submitted 2019-11-07; First posted 2019-11-12 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Term Pregnancy; Doppler Parameters; Induction of Labor; Fetal Complications
Keywords: term pregnancy; Doppler parameters; Cerebroplacental ratio; Induction of labor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Pregnant women with CPR value below 1, based on Doppler indices assessment
  Interventions: Diagnostic Test: Doppler flow indices assessment
- Group 2: Pregnant women with CPR value equal to or above 1, based on Doppler indices assessment
  Interventions: Diagnostic Test: Doppler flow indices assessment

INTERVENTIONS:
Diagnostic Test: Doppler flow indices assessment — Doppler flow indices, UA-PI, MCA-PI and CPR values, assessment performed prior to induction of labor

SUMMARY:
Term pregnancies within their 37-41 gestational week, who were planned to undergo induction of labor, were included in the study. Prior to initiation of the induction of labor, all included pregnant women underwent an assessment of Doppler flow indices, which included fetal umblical artery PI (pulsatility index) and fetal middle cerebral artery (MCA:Middle cerebral arter) PI. Cerebroplacental Ratio (CPR) was calculated by dividing MCA PI value to umbilical artery PI (MCA PI/UA PI=CPR).Included pregnant women were categorized as Group 1 and Group 2, which comprised of those with CPR value below 1.0 and above 1.0, respectively. Route of delivery and fetal complications, described as umbilical cord pH<7.20, APGAR score at 5 minutes <7, meconium aspiration syndrome, newborn intensive care unit admission, neonatal sepsis and neonatal death.

DETAILED DESCRIPTION:
Term pregnancies within their 37-41 gestational week, who were planned to undergo induction of labor, were included in the study. Prior to initiation of the induction of labor, all included pregnant women underwent an assessment of Doppler flow indices, which included fetal umblical artery PI (pulsatility index) and fetal middle cerebral artery (MCA:Middle cerebral arter) PI. Cerebroplacental Ratio (CPR) was calculated by dividing MCA PI value to umbilical artery PI (MCA PI/UA PI=CPR).Included pregnant women were categorized as Group 1 and Group 2, which comprised of those with CPR value below 1.0 and above 1.0, respectively. All women who were considered appropriate for induction of labor were performed an pelvic examination and their Bishop scores were calculated. Those with a Bishop score equal to or below 5 were included in the study. Vaginal misoprostol (prostoglandin E1, 25 mcg) and dinoproston (prostoglandin E2, 10 mg) were used for induction of labor. Repeat doses were implemented in case of insufficient cervical ripening. Oxytocin was not used at the initial stages of labour, while it was used at the latter stages when necessary.

Route of delivery and fetal complications, described as umbilical cord pH<7.20, APGAR score at 5 minutes <7, meconium aspiration syndrome, newborn intensive care unit admission, neonatal sepsis and neonatal death.

ELIGIBILITY:
Inclusion Criteria:

* Term pregnancies between 37 and 41 gestational weeks Pregnancies destined to induction of labor

Exclusion Criteria:

* history of uterine scar, nonverteks presentation, multiple pregnancies, use of vacuum of forceps at delivery, shoulder dystocia, confirmed fetal structural or chromosomal anomalies

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Term pregnancies within their 37-41 gestational week, who were planned to undergo induction of labor, were included in the study. Prior to initiation of the induction of labor, all included pregnant women underwent an assessment of Doppler flow indices, which included fetal umblical artery PI (pulsatility index) and fetal middle cerebral artery (MCA:Middle cerebral arter) PI.
Sampling Method: Non-Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Umblical arter pH | Within 1-3 minutes following delivery
  Umbilical cord blood sampling just after the delivery of the newborn and pH measurement
APGAR score at 5 minutes | Postpartum 5 minutes
  APGAR score determined by the pediatrician at postpartum 5 minutes
Meconium aspiration syndrome | Within postpartum two weeks
  Meconium aspiration syndrome diagnosed by the pediatrician, either clinically or by thorax X-ray film.
Newborn intensive care unit administration | Within postpartum 1 month period
  Newborn intensive care unit administration, due to a variety of conditions, which were established by pediatrician
Neonatal sepsis | Within postpartum 1 month period
  Neonatal sepsis diagnosed by the pediatrician
Neonatal death | Within postpartum 1 month period
  Neonatal death

SECONDARY OUTCOMES:
Route of delivery | At the time of delivery
  Route of delivery, either vaginally or by cesarean section

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medeniyet University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP